CLINICAL TRIAL: NCT01611077
Title: Efficacy and Safety of a Sequential Therapy Change From Candesartan 32 mg to the Fixed Combination of Olmesartan 40 mg/Amlodipine 10 mg in Patients With Poorly Controlled Moderate Hypertension - an Open Phase IV Trial
Brief Title: Efficacy and Safety of a Therapy Change From Candesartan 32 mg to Fixed Combination of Olmesartan 40 mg/Amlodipine 10 mg
Acronym: Sevicontrol-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sevicontrol-2
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Olmesartan Medoxomil; olmesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): Candesartan 16 mg tablets p. o. once daily for 14 days, 32 mg tablets once daily for 28 days, then olmesartan 40 mg tablets once daily for 42 days, then olmesartan/amlodipine 40/5 mg tablets once daily for 14 days, then olmesartan/amlodipine 40/10 mg tablets once daily for 28 days
  Interventions: Drug: Candesartan cilexetil; Drug: Olmesartan medoxomil; Drug: Olmesartan/amlodipine

INTERVENTIONS:
Drug: Candesartan cilexetil — Candesartan 16 mg tablets p. o. once daily for 14 days, 32 mg tablets once daily for 28 days
  Other Names: Atacand
Drug: Olmesartan medoxomil — Switch to olmesartan 40 mg tablets once daily for 42 days,
  Other Names: Olmetec
Drug: Olmesartan/amlodipine — then switch to olmesartan/amlodipine 40/5 mg tablets once daily for 14 days, then olmesartan/amlodipine 40/10 mg tablets once daily for 28 days
  Other Names: Sevikar (r)

SUMMARY:
The investigators want to find out if a treatment with a new combination of two different antihypertensive drugs (olmesartan and amlodipine) in one tablet in patients with moderately elevated blood pressure is more effective than treatment with just one substance (candesartan). All antihypertensive treatment will be ceased for two weeks to achieve comparable baseline conditions. Treatment is then started with the single substance. After six weeks, therapy is changed to another single substance and after a further six weeks, to the fixed combination tablet. Blood pressure is determined by office measurements taken by the doctor and via long-term ambulatory blood pressure monitoring (ABPM). Participants may be male or female and must be over 18 years of age.

DETAILED DESCRIPTION:
SEVICONTROL-2:

Efficacy and Safety of a sequential therapy change from Candesartan 32 mg to the fixed combination of olmesartan 40 mg/amlodipine 10 mg in patients with poorly controlled moderate hypertension - an open phase IV trial

ELIGIBILITY:
Inclusion Criteria:

* male or female patients >= 18 years of age
* essential hypertension, i. e. systolic office bp >= 140 mmHg for pre-treated patients or >= 160 mmHg for untreated patients at screening visit and >= 160 mmHg at end of wash-out
* signed IC

Exclusion Criteria:

* systolic office bp > 180 mm Hg at screening visit
* known hypertensive retinopathy GIII or IV
* recent (< 4 weeks ago) myocardial infarction or indication for coronary or peripheral revascularisation
* type I diabetes or poorly controlled (HbA1c >= 8) type II diabetes
* chronic heart failure NYHA III or IV
* prior stroke or TIA
* creatinine clearance < 60 ml/min or condition after kidney transplant
* moderately or severely impaired liver function (ALT or AST or bilirubin more than double normal value)
* women of childbearing potential without highly effective contraception, pregnant or breastfeeding women
* concomitant therapy with lithium
* hemodynamically relevant mitral or aortic valve stenosis (>= II°) or hypertrophic obstructive cardiomyopathy
* concomitant therapy with strong CYP3A4 inhibitors or inductors
* african patients
* concomitant severe psychiatric condition that might impair proper intake of study medication
* life expectancy < 6 months
* night shift workers
* known other mandatory indication for treatment with antihypertensive medications
* parallel participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic daytime mean ABPM (long-term ambulatory blood pressure monitoring) values | ABPM will be performed after 6 weeks treatment with each of the different therapy regimes.
  After six weeks therapy with a monotherapy with olmesartan 40 mg and further six weeks treatment with a fixed combination of olmesartan 40 mg and amlodipine 10 mg compared to previous monotherapy with candesartan.

SECONDARY OUTCOMES:
Change in systolic/diastolic office blood pressure and mean values (night-time and 24 hr for systolic bp and day-time, night-time and 24 hr for diastolic bp) | after 6 and 12 weeks
  from candesartan to olmesartan 40 mg and then to a fixed combination of olmesartan 40 mg and amlodipine 10 mg.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Lüders, Dr.med., Principal Investigator — St.-Josefs-Hospital Cloppenburg
Locations (11):
- Germany (11):
  - Praxis Dr. Reimer, Anderbeck
  - Praxis Dr. Heinz, Bergisch Gladbach
  - Praxis Dr. Zemmrich, Berlin
  - St.-Josefs-Hospital, Cloppenburg
  - Praxis Dr. Pohl, Dresden
  - Praxis Dr. Koßler-Wiesweg, Essen
  - Praxis Dr. Rövenich, Frankfurt
  - Praxis Dr. Strzata, Kapellendorf
  - Praxis Dr. Paschmionka, Leipzig
  - Praxis Dr. Pitule, Ludwigshafen
  - Praxis Dr. Loddo, Rastede

IPD SHARING:
Plan to Share IPD: Undecided